CLINICAL TRIAL: NCT02732574
Title: The Effectiveness of Oscillating Positive Expiratory Pressure (OPEP) Therapy in High Risk Patients Following Cardiac Surgery Surgery: A Randomized Clinical Trial
Brief Title: Oscillating Positive Expiratory Pressure (OPEP) Therapy in High Risk Patients Following Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Philip Jones, Associate Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPEP-2016
Record Dates: First submitted 2016-03-27; First posted 2016-04-08 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass Grafting; Chronic Obstructive Pulmonary Disease (COPD); Older Adults; Postoperative Pulmonary Complications
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPEP Device Treatment (Experimental): Patients randomized to OPEP will receive the device on postoperative day (POD) 1 or day of extubation, whichever comes first. Patients will be seen on POD #1 by a blinded physiotherapist (PT) for mobility and education on supported coughing. The OPEP device group will also be instructed to complete 15 breaths twice per waking hour in a seated position and receive education on proper use of the device. The OPEP device will be set to the highest pressure setting unless deemed inappropriate by the PT, at which time the most appropriate pressure setting will be selected and then increased daily until the OPEP device is set to the highest pressure setting by POD #3 if able. The PT will reassess the patients on POD 2 and 3 to assess for proper technique and continued use of the device, as well as usual care. Patients will use the OPEP device up to POD#5 pressure settings and compliance will be recorded and measure by use of a daily log.
  Interventions: Device: Oscilatory Positive Expiratory Pressure (OPEP) device
- SHAM Device (Sham Comparator): Patients randomized to the sham treatment will receive the sham device on postoperative day (POD) 1 or day of extubation, whichever comes first. Patients will be seen on POD #1 by a blinded physiotherapist (PT) for mobility and education on supported coughing. The sham group will also be instructed to complete 15 breaths twice per waking hour in a seated position and receive education on proper use of the device. The sham device is identical in exterior appearance to the OPEP device but does not contain the internal mechanism providing expiratory pressure. As such, the device will be set to the highest setting and will not need to be adjusted at all for patient tolerance. The PT will reassess the patients on POD 2 and 3 to assess for proper technique and continued use of the device, as well as usual care. Patients will use the OPEP device up to POD#5 pressure settings and compliance will be recorded and measure by use of a daily log.
  Interventions: Device: SHAM Device Group

INTERVENTIONS:
Device: Oscilatory Positive Expiratory Pressure (OPEP) device — OPEP devices will be set to the highest pressure setting tolerated on POD #1. If the highest pressure setting is not achieved on POD#1, the PT will increase the pressure daily with the aim to achieve the highest pressure setting as soon as tolerated by the patient or POD#3, whichever comes first. Patients will be instructed to complete 15 breaths in a seated position with the OPEP device twice per waking hour. This will occur in addition to usual care.
  Other Names: Aerobika
  Arms: OPEP Device Treatment
Device: SHAM Device Group — SHAM devices will be provided to patients on POD #1 and set to the highest pressure setting externally, however no positive expiratory pressure will be provided as the internal pressure regulating mechanism has been removed. Patients will be instructed to complete 15 breaths in a seated position with the sham device twice per waking hour. This will occur in addition to usual care.
  Arms: SHAM Device

SUMMARY:
Respiratory dysfunction following cardiac surgery is well documented and due in part to the location of the incision and nature of the surgery. Post-operative pulmonary complications (PPCs) remain a significant problem following cardiac surgery, sometimes causing prolonged length of stay in hospital as well as increased morbidity and mortality; with the greater risk to older adults and individuals with obstructive lung disease. Positive expiratory pressure (PEP) therapy is thought to increase lung volumes and facilitate secretion clearance. The purpose of this study is to investigate whether the addition of oscillating PEP therapy to standard postoperative treatment is more effective in decreasing the incidence of PPCs and increasing functional capacity at time of discharge in 'high risk' patients undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
Respiratory dysfunction following cardiac surgery is well documented and due in part to the location of the incision and nature of the surgery (Weissman, 2000; Garcia-Delgado M, et al., 2014). Patients undergoing cardiac surgery are at an increased risk of postoperative pulmonary complications including hypoxemia, atelectasis, and pneumonia (Weissman, 2000; Garcia-Delgado M, et al., 2014; O'Donohue WJ, 1992); with an increased risk in older individuals and individuals with obstructive lung disease (Crowe & Bradley, 1997; Weissman 2000; Jensen et al., 2007). Standard postoperative care includes early mobility and deep breathing and coughing (DB&C) (Stiller K, et al., 1995; Johnson D., et al., 1996) usually initiated within the first 24 hours following surgery. Although standard care is sufficient in some instances, postoperative pulmonary complications (PPCs) remain a significant problem following cardiac surgery and can cause prolonged length of stay in the hospital and an increase in morbidity and mortality (Weissman, 2000; Garcia-Delgado M, et al., 2014) in a significant number of patients. Positive expiratory pressure (PEP) therapy is thought to increase lung volumes and facilitate secretion clearance in many populations (Orman J & Wasterdahl E, 2009) and has been shown to be particularly effective in individuals with obstructive lung disease (Bott et al ., 2009). In consideration of the well documented respiratory dysfunction observed following cardiac surgery, PEP therapy may serve as a promising treatment in facilitating recovery in older, 'higher risk' individuals following elective cardiac surgery. Thus, the purpose of this study is to investigate whether the addition of oscillating PEP therapy is more effective than standard treatment alone in improving functional status at time of discharge, as well as decreasing oxygen requirements and the incidence of postoperative pulmonary complications (e.g., pneumonia, atelectasis, pneumothorax, pleural effusions) in 'high risk' patients undergoing elective cardiac surgery.

Participants will be recruited from London Health Sciences Centre in London Ontario. Patients deciding to proceed with elective cardiac surgery will be screened in the surgeon's office, pre-admission clinic or the 6-inpatient ward for eligibility to participate in the study and provided with a letter of information. Each patient will be required to provide written consent in order to participate in this study. The study will be approved by the Health Sciences Research Ethics Board at Western University. Patients who have consented to participation in the study will be seen by the research coordinator at the patient's pre-operative clinic appointment where the research coordinator will explain the purpose and nature of the study and obtain written informed consent. Also, at that time, patient demographic information will be collected, as well as baseline data of chest x-ray (CXR) and a six minute walk test (6MWT). Pre-operative 6MWTs will be performed on a standardized 30 meter track in the basement of University Hospital and will comply with the American Thoracic Society Guidelines (2002). Patients enrolled in the study will be randomized to one of two groups on the day of their surgery; OPEP treatment or sham treatment group. On the day of surgery or post-operative day (POD) 1, the research coordinator will bring the device (OPEP or sham depending on randomization) to the patient's room. The sham devices have been manufactured to be externally identical to the OPEP devices allowing for patient blinding, however the sham devices do not contain the internal mechanisms provided expiratory pressure. All patients (sham or OPEP) will be seen by a physiotherapist on the day of extubation and receive instructions on how to properly use the device, in addition to receiving standard post-operative care. Patients will be instructed to set the resistance on the device to the highest setting and perform up to 15 breaths in the sitting position at least twice per waking hour. The resistance and number of repetitions may be decreased to adjust for patient tolerance as deemed appropriate by the treating physiotherapist. Compliance will be measured through a log book completed by the patient and/or their family. Patients will be reassessed by a physiotherapist on POD #2 and #3 to ensure proper technique and compliance with the device. All patients will continue to receive standard care each day as per the clinical pathway and may receive additional cardiorespiratory PT techniques as deemed necessary by the PT. Patients will be instructed to continue with OPEP treatments (sham or OPEP) as described until POD #5. Outcome assessment will be conducted by a blinded assessor. The outcomes and timing of outcome assessment is described in the outcome measures section and will terminate on POD #7 or discharge from hospital, whichever occurs first. If patients require continuous positive airway pressure (CPAP), bilevel positive airway pressure (BiPAP), or reintubation during this period, they will be instructed to stop using their OPEP device and outcome assessment will occur only until POD#7.

ELIGIBILITY:
Undergoing elective or urgent coronary artery bypass grafting (CABG) surgery at London Health Sciences Centre and satisfying the following criteria:

Inclusion Criteria:

* CABG surgery or CABG-one valve (mitral or aortic) surgery (including conventional sternotomy on cardiopulmonary bypass, minimally-invasive and off-pump surgery)
* Age >= 60 years
* Documentation of at least one of the following: (pre-operative fraction of expired volume in one second (FEV1) of less than 70% predicted), (pre-operative FEV1/forced vital capacity (FVC) of less than 80%), or (on any daily usage of inhaled anti-cholinergic, beta2-agonist, or corticosteroid)
* New York Heart Association (NYHA) ≥ 2

Exclusion criteria:

* Patients not meeting inclusion for high risk surgical candidate
* Unable/unwilling to provide written informed consent
* Patients undergoing emergent cardiac surgery
* Untreated postoperative pneumothorax
* Patients on home CPAP or BiPAP therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT) Distance (meters) | Postoperative day 5
  A 6MWT will be conducted as per American Thoracic Society guidelines in a designated hallway in the basement of university hospital or a corridor outside the cardiac surgery recovery unit. The tests will be conducted by a blinded assessor pre-operatively and on Postoperative day 5 or day of discharge, whichever comes first. Distance walked in meters will be recorded.

SECONDARY OUTCOMES:
Total duration of oxygen therapy | Time of tracheal extubation to Postoperative day 7
  Cumulative duration of oxygen therapy will be tracked and recorded for all patients, tracked from time of extubation until Postoperative day 7 or discharge, whichever comes first.
Total exposure to oxygen therapy | From tracheal extubation until Postoperative day 7
  The cumulative exposure to oxygen post-extubation will be tracked by calculating an area under the dose-time curve for oxygen usage, tracked from time of extubation until Postoperative day 7 or discharge, whichever comes first..
Number of cycles between room air and oxygen supplementation | From tracheal extubation until Postoperative day 7
  Each time someone goes from room air to back on oxygen, this is a setback, and we will count this one 'cycle', tracked from time of extubation until Postoperative day 7 or discharge, whichever comes first..
Incidence of postoperative pulmonary complications (PPCs) as determined by CXR interpretation | Postoperative days 1 and 4
  Incidence of PPCs will be assessed by a blinded assessor. PPCs will include:
  * pneumonia/consolidation
  * atelectasis
  * pleural effusions
  * pulmonary edema
  * pneumothorax.
  Presence of each PPC will be expressed as a 3 point score: 0= absent, 1=mild (not likely clinically relevant), 2 = moderate to severe (likely clinically relevant).
Intensive Care Unit (ICU) length of stay (LOS) | Through study completion
  time from admission to ICU (time 0) until actual discharge from ICU
Hospital LOS | Through study completion
  Time from admission to ICU until actual discharge from hospital
All-cause 30-day mortality | Up to and including the 30th post-operative day
  This will be determined by hospital records, a phone call to family physician (if available) or by phone call to patient or substitute decision maker.

OTHER OUTCOMES:
Number of sham or OPEP device uses | Days 1 through 5
CPAP usage | Up to postoperative day 7
  Any patient who post-extubation requires CPAP therapy.
BiPAP usage | Up to postoperative day 7
  Any patient who post-extubation requires BiPAP therapy.
Re-intubation | Up to postoperative day 7
  Any patient who post-extubation requires re-intubation of the trachea.
Borg shortness of breath scale | Through study completion
  During the postoperative six-minute walk test (on postoperative day 5 or discharge date, whichever comes first)
Fatigue scale while performing six minute walk test | Through study completion
  The patient will assess their overall level of fatigue during the 6-min walk test on numeric rating scale (0 - not at all fatigued, 10 - maximally fatigued). During postoperative six minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jones, MD, MSc (Clinical Trials), Principal Investigator — Western University, Canada
Locations (1):
- University Hospital - London Health Sciences Centre, London, Ontario, Canada